CLINICAL TRIAL: NCT03230383
Title: A Phase 1, Randomized, Double-blind, Placebo-controlled Study To Assess The Safety, Tolerability, And Pharmacokinetics Of Multiple Escalating Oral Doses Of PF-06865571 In Healthy, Including Overweight And Obese, Adult Subjects
Brief Title: A Study To Assess The Safety, Tolerability, And Pharmacokinetics (PK) Of Multiple Doses Of PF-06865571 In Healthy, Including Overweight And Obese, Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Basic Science
Other Study IDs: C2541002; 2017-001649-28 (EudraCT Number)
Record Dates: First submitted 2017-07-24; First posted 2017-07-26 (Actual); Last update posted 2018-05-23 (Actual); Status verified 2018-05

CONDITIONS: Healthy Subjects
MeSH Terms: interventions — ervogastat

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Cohort 1_90mg and Matching Placebo (Experimental)
  Interventions: Drug: PF-06865571; Drug: Placebo
- Cohort 2_300mg and Matching Placebo (Experimental)
  Interventions: Drug: PF-06865571; Drug: Placebo
- Cohort 3_900mg and Matching Placebo (Experimental)
  Interventions: Drug: PF-06865571; Drug: Placebo
- Cohort 4_1800mg and Matching Placebo (Experimental)
  Interventions: Drug: PF-06865571; Drug: Placebo
- Cohort 5_3000mg and Matching Placebo (Experimental)
  Interventions: Drug: PF-06865571; Drug: Placebo
- Optional Cohort 6_TBD mg and Matching Placebo (Experimental)
  Interventions: Drug: PF-06865571; Drug: Placebo
- Optional Cohort 7_TBD mg and Matching Placebo (Experimental)
  Interventions: Drug: PF-06865571; Drug: Placebo

INTERVENTIONS:
Drug: PF-06865571 — Multiple ascending dose of PF-06865571 as extemporaneously prepared suspension for 14 consecutive days with total daily dose of 90mg, 300mg, 900mg, 1800mg, 3000mg and TBD.
  Arms: Cohort 1_90mg and Matching Placebo
Drug: PF-06865571 — Multiple ascending dose of PF-06865571 as extemporaneously prepared suspension for 14 consecutive days with total daily dose of 90mg, 300mg, 900mg, 1800mg, 3000mg and TBD.
  Arms: Cohort 2_300mg and Matching Placebo
Drug: PF-06865571 — Multiple ascending dose of PF-06865571 as extemporaneously prepared suspension for 14 consecutive days with total daily dose of 90mg, 300mg, 900mg, 1800mg, 3000mg and TBD.
  Arms: Cohort 3_900mg and Matching Placebo
Drug: PF-06865571 — Multiple ascending dose of PF-06865571 as extemporaneously prepared suspension for 14 consecutive days with total daily dose of 90mg, 300mg, 900mg, 1800mg, 3000mg and TBD.
  Arms: Cohort 4_1800mg and Matching Placebo
Drug: PF-06865571 — Multiple ascending dose of PF-06865571 as extemporaneously prepared suspension for 14 consecutive days with total daily dose of 90mg, 300mg, 900mg, 1800mg, 3000mg and TBD.
  Arms: Cohort 5_3000mg and Matching Placebo
Drug: PF-06865571 — Multiple ascending dose of PF-06865571 as extemporaneously prepared suspension for 14 consecutive days with total daily dose of 90mg, 300mg, 900mg, 1800mg, 3000mg and TBD.
  Arms: Optional Cohort 6_TBD mg and Matching Placebo
Drug: PF-06865571 — Multiple ascending dose of PF-06865571 as extemporaneously prepared suspension for 14 consecutive days with total daily dose of 90mg, 300mg, 900mg, 1800mg, 3000mg and TBD.
  Arms: Optional Cohort 7_TBD mg and Matching Placebo
Drug: Placebo — Matching Placebo for PF-06865571 for each cohort.

SUMMARY:
This will be an investigator- and subject-blinded (sponsor open), randomized, placebo controlled, sequential, ascending, multiple oral dose study, with 5 planned cohorts (optional sixth and seventh cohorts). A total of approximately 50 (if 5 cohorts), 60 (if 6 cohorts), and up to 70 (if 7 cohorts) subjects will be randomized in this study. Subjects in each cohort will be randomized to receive PF-06865571 or matching placebo with approximately 10 subjects dosed in each cohort.

For a given subject in any cohort, the total study duration from screening to follow-up phone call will be between approximately 7 to 11 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males and female of non-childbearing potential;
* Age of 18-55, inclusive;
* Body Mass Index 22.5 to 35.4 kg/m2, inclusive;
* Body weight greater than 50 kg;
* Not on any prescription or non-prescription drugs within 7 days or 5 half-lives prior to first dose.

Exclusion Criteria:

* Evidence of history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including drug allergises, but excluding untreated, asymptomatic, seasonal allergies at time of dosing);
* Subjects with fasting LDL-C level >190 mg/dL following an overnight fast of at least 10 hours, at the Screening visit, confirmed by a single repeat, if deemed necessary.
* Subjects with fasting TG level >400 mg/dL following an overnight fast of at least 10 hours, at the Screening visit, confirmed by a single repeat, if deemed necessary.
* Any condition possibly affecting drug absorption (eg, gastrectomy).
* A positive urine drug test.
* History of regular alcohol consumption exceeding 7 drinks/week for female subjects or 14 drinks/week for male subjects (1 drink = 5 ounces [150 mL] of wine or 12 ounces [360 mL] of beer or 1.5 ounces [45 mL] of hard liquor) within 6 months before screening.
* Treatment with an investigational drug within 30 days (or as determined by the local requirement) or 5 half lives preceding the first dose of investigational product (whichever is longer).
* Use of tobacco- or nicotine-containing products in excess of the equivalent of 5 cigarettes per day or 2 chews of tobacco per day.
* Pregnant female subjects; breastfeeding female subjects; male subjects with partners currently pregnant; fertile male subjects who are unwilling or unable to use a highly effective method of contraception as outlined in this protocol for the duration of the study and for at least 28 days after the last dose of investigational product.
* Unwilling or unable to comply with the criteria in the Lifestyle Requirements section of this protocol.
* Other acute or chronic medical or psychiatric condition including recent (within the past year) or active suicidal ideation or behavior or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the subject inappropriate for entry into this study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2018-05-03 (Actual); Study Completion 2018-05-03 (Actual)

PRIMARY OUTCOMES:
Number of subjects with adverse events (AEs) | Baseline up to 35 days after last dose of study medication
  Number of participants with reported adverse events
Number of subjects with laboratory tests findings of potential clinical importance | Baseline (Day 0) up to 24 days after last dose of study medication
  Number of participants with potentially clinically important laboratory test findings
Number of subjects with electrocardiogram (ECG) findings of potential clinical importance | Baseline (Day 0) up to 24 days after last dose of study medication
  Number of participants with potentially clinically important ECG findings
Number of subjects with vital signs findings of potential clinical importance | Baseline (Day 0) up to 24 days after last dose of study medication
  Number of participants with potentially clinically important vital sign measurements

SECONDARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) for PF-06865571 | 0, 0.5, 1, 2, 3, 4, 6, 8, 10, 12 hour post dose on Days 1, 7, and 14
AUCtau for PF-06865571 | 0, 0.5, 1, 2, 3, 4, 6, 8, 10, 12 hour post dose on Days 1, 7, and 14
  Area under the concentration-time curve calculated by linear trapezoidal rule from time zero to the end of the dosing interval (i.e., 24 h) at steady state.
Time to Reach Maximum Observed Concentration for PF-06865571 | 0, 0.5, 1, 2, 3, 4, 6, 8, 10, 12 hour post dose on Days 1, 7, and 14
  Time to Reach Maximum Observed Plasma Concentration (Tmax)
Dose normalized Cmax for PF-06865571 | 0, 0.5, 1, 2, 3, 4, 6, 8, 10, 12 hour post dose on Days 1, 7, and 14
  Following log-transformation, dose normalized Cmax will be analysed using a mixed model appropriate to the study design.
Amount of unchanged drug recovered in urine during the dosing interval (Aetau) for PF-06865571 | 0, 0.5, 1, 2, 3, 4, 6, 8, 10, 12 hour post dose on Day 14
  Sum of [urine concentration * sample volume] for each collection over the dosing interval
Percent of dose recovered in urine as unchanged drug (Aetau %) for PF-06865571 | 0, 0.5, 1, 2, 3, 4, 6, 8, 10, 12 hour post dose on Day 14
  100* Aetau/Dose
Renal clearance (CLr) for PF-06865571 | 0, 0.5, 1, 2, 3, 4, 6, 8, 10, 12 hour post dose on Day 14
  Aetau/AUCtau

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (2):
- Pfizer New Haven Clinical Research Unit, New Haven, Connecticut, United States
- Pfizer Clinical Research Unit, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No
Information relating to our policy on data sharing and the process for requesting data can be found at the following link: http://www.pfizer.com/research/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Amin NB, Saxena AR, Somayaji V, Dullea R. Inhibition of Diacylglycerol Acyltransferase 2 Versus Diacylglycerol Acyltransferase 1: Potential Therapeutic Implications of Pharmacology. Clin Ther. 2023 Jan;45(1):55-70. doi: 10.1016/j.clinthera.2022.12.008. Epub 2023 Jan 21. PMID 36690550
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=C2541002&StudyName=A+Phase+1%2C+Randomized%2C+Double+Blind%2C+Placebo+Controlled+Study+To+Assess+The+Safety%2C+Tolerability%2C+And+Pharmacokinetics+Of+Multiple+Escalating+Oral+Doses+Of+Pf+06865571+In+Otherwise+Healthy%2C+Adult+Subjects
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=C2541002&StudyName=A+Phase+1%2C+Randomized%2C+Double-blind%2C+Placebo-controlled+Study+To+Assess+The+Safety%2C+Tolerability%2C+And+Pharmacokinetics+Of+Multiple+Escalating+Oral+Doses+Of+Pf-06865571+In+Healthy%2C+Including+Overweight+And+Obese%2C+Adult+Subjects